CLINICAL TRIAL: NCT03979248
Title: An Open-Label, Single-Sequence Study to Investigate the Effects of Gastric Acid Suppression by Rabeprazole on the Pharmacokinetics of BMS-986165 in Healthy Participants
Brief Title: A Study to Investigate the Effects of Gastric Acid Suppression by Rabeprazole and BMS-986165 on How Fast and Complete The Drug is Absorbed Into the Body of Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM011-090; 2019-001193-28 (EudraCT Number)
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Healthy
MeSH Terms: interventions — deucravacitinib; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMS-986165 + Rabeprazole (Experimental)
  Interventions: Drug: BMS-986165; Drug: Rabeprazole

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days.
Drug: Rabeprazole — Specified dose on specified days.

SUMMARY:
The purpose of this study is to evaluate the effects of stomach acid suppression by rabeprazole and BMS-986165 on how fast and complete the drug is absorbed into the body of healthy participants.

ELIGIBILITY:
Inclusion Criteria

* Healthy participant, as determined by medical history, physical examination, ECGs, and clinical laboratory determinations
* Body mass index of 18.0 kilogram per meter square (kg/m^2) to 32.0 kg/m^2
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) greater than (>) 80 milliliter per minute per 1.732 meter square (mL/min/1.732 m^2)

Exclusion Criteria:

* Any major surgery within 4 weeks of study drug administration
* Use of any prescription drugs or over-the-counter acid controllers
* Positive urine screen for drugs of abuse, alcohol, or cotinine
* History of allergy to BMS-986165, rabeprazole, or related compounds

Other protocol inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of BMS-986165 | Day 1 and Day 9
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-T]) of BMS-986165 | Day 1 and Day 9
Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC[INF]) of BMS-986165 | Day 1 and Day 9

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to Day 12
Percentage of Participants with Clinical Laboratory Values, Vital Signs, and Electrocardiograms (ECGs) | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Netherlands, Groningen, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm